CLINICAL TRIAL: NCT02921594
Title: Comparison of Vanguard XP and Vanguard CR Total Knee Arthroplasties: A Cross Sectional Pilot Study Evaluating Intraarticular Kinematics and Standing Balance by Dynamic Fluoroscopy and Force Plate Examination
Brief Title: Kinematic Comparison of Vanguard XP and Vanguard CR Total Knee Arthroplasties
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: NCT02921594 was not a RCT but a secondary pilot study designed to establish a fluoroscopic test-set up on 10 selected patients from another RCT.
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Anders Troelsen, Professor, MD, PhD, dr.med, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XPvsCR_Fluoroscopi_v.1.0
Record Dates: First submitted 2016-09-26; First posted 2016-10-03 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Total knee arthroplasty with Vanguard XP (Active Comparator): The new Vanguard XP Total knee arthroplasty system is a further development of the Vanguard TKA. The new Vanguard XP system both cruciate ligaments are preserved.
  Interventions: Device: Total knee arthroplasty with Vanguard XP; Device: Total knee arthroplasty with Vanguard CR
- Total knee arthroplasty with Vanguard CR (Active Comparator): Total knee arthroplasty system without preservation of the anterior cruciate ligament
  Interventions: Device: Total knee arthroplasty with Vanguard XP; Device: Total knee arthroplasty with Vanguard CR

INTERVENTIONS:
Device: Total knee arthroplasty with Vanguard XP
Device: Total knee arthroplasty with Vanguard CR

SUMMARY:
Primary: The primary objective of this pilot study is to compare the intraarticular kinematics by fluoroscopy of Vanguard XP to that of Vanguard CR.

Secondary: The secondary objective of this pilot study is to compare the standing balance by force plate of patients with the Vanguard XP prosthesis to those who have Vanguard CR prosthesis. Furthermore, we wish to assess isometric quadriceps muscle strength in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Participant in the XP vs. CR study (inherited traits from study inclusion)
* Overall healthy. Have attended standard physiotherapy after unilateral total knee replacement
* Are able to perform the tasks
* Excellent clinical scores (Oxford Knee Score above 39 at 1 year follow up)

Exclusion Criteria:

* Knee pain above 20 on a 0-100 visual analogue scale
* Any clinical relevant pain from adjacent joints
* Active Knee flexion below 100
* Signs of implant migration, loosening, and implant mal-alignment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2017-03 (Estimated); Study Completion 2018-08-16 (Actual)

PRIMARY OUTCOMES:
Anterior-posterior translation of the femoral component with respect to the tibia component | at least one year post surgery
  Group mean in millimeters (mm)
Axial rotation of the femoral component with respect to the tibia component | at least one year post surgery
  Group mean in degrees (°)

SECONDARY OUTCOMES:
Traveled distance of center of pressure | at least one year post surgery
  Group mean in centimeters (cm)
Velocity of center of pressure | at least one year post surgery
  Group mean in mm/second
Rambling-trembling distance | at least one year post surgery
  Group mean in mm
Isometric quadriceps muscle strength | at least one year post surgery
  Group mean in newton meter pr. kilograms weight (Nm/kg)

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Orthopaedic Surgery, Copenhagen University Hospital Hvidovre, Hvidovre, Denmark